CLINICAL TRIAL: NCT05637541
Title: A Randomized, Double-blind, Placebo-controlled and Multicenter Phase Ⅱ Clinical Trials To Evaluate the Safety, Efficacy and Pharmacokinetics of GST-HG141 Tablets in Treated Chronic Hepatitis B (CHB) Patients With Low Viremia
Brief Title: Evaluation of The Safety, Efficacy and Pharmacokinetic Characteristics of GST-HG141 Tablets
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Akeylink Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GST-HG141-Ⅱ-02
Record Dates: First submitted 2022-11-24; First posted 2022-12-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2024-08

CONDITIONS: Chronic Hepatitis b
Keywords: Chronic Hepatitis b
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-dose group (Experimental): Drug 1 is a vial of 130 tablets of the experimental drug, and drug 2 is a vial of 130 tablets of the placebo
  Interventions: Drug: GST-HG141
- High-dose group (Experimental): Drug 1 and 2 are each a vial of 130 tablets of the experimental drug
  Interventions: Drug: GST-HG141
- Placebo group (Placebo Comparator): Drug 1 and drug 2 are each a vial of 130 tablets of the placebo
  Interventions: Drug: GST-HG141

INTERVENTIONS:
Drug: GST-HG141 — The trial consisted of a low-dose group and a high-dose group, each of which was 50mg bid and 100mg bid for 12 or 24 weeks of treatment

SUMMARY:
A Randomized, Double-blind, Placebo-controlled and Multicenter Phase Ⅱ Clinical Trials To Evaluate the Safety, Efficacy and Pharmacokinetics of GST-HG141 Tablets in Treated Chronic Hepatitis B (CHB) Patients With Low Viremia.

DETAILED DESCRIPTION:
This study was a multicenter, randomized, double-blind, placebo-controlled phase II clinical trial to evaluate the efficacy and safety of different doses of GST-HG141 in treated CHB patients with low viremia.

A total of 90 CHB patients with low viremia after hepatitis B antiviral therapy were enrolled in this study, and they were divided into three groups, 30 cases in each group. Screening of eligible subjects, according to the proportion were randomly assigned to: GST - HG141 low dose group, the GST - HG141 high dose group and the placebo group.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent before the trial and fully understand the content, process and possible adverse reactions of the trial;
2. Ability to complete research in accordance with test plan requirements;
3. Subjects (including partners) are willing to take effective pregnancy avoidance measures within 28 days after screening to the last study drug administration;
4. Male and female subjects aged between 18 and 70 years old (both inclusive);
5. The weight of male subjects shall not be less than 50kg and that of female subjects shall not be less than 45kg. Body mass index (BMI) = body weight (kg) / height 2 (M2), and the body mass index is within the range of 18-35 kg / m2 (including the critical value);
6. Have been taking a nucleoside analogue (entecavir [ETV], tenofovir dipiroxide fumarate [TDF], or profotenofovir [TAF]) for 1 to 3 years, were receiving treatment at the time of screening and agreed to receive the treatment offered in this study during the study;
7. Serum HBV DNA could be detected by high-sensitivity PCR with a dose of 20 IU/ ml < HBV DNA < 2000 IU/mL;
8. Screening, ALT ≤ 5 x ULN and liver stiffness testing (LSM) meet the following requirements: ALT≤ 2 x ULN, LSM≤10.6 kPa; Or 2 x ULN≤ ALT≤ 5×ULN ，LSM< 12.4 kPa.

Exclusion Criteria:

1. Patients with a history of allergy or suspected allergy to the active ingredient or excipients of the drug under study;
2. Concomitant use of an inhibitor, inducer, or substrate of the cytochrome P450 enzyme 3A4 isoenzyme (CYP3A4) within 28 days before screening；
3. Patients with systemic use of immunosuppressants, immunomodulators (excluding interferon) and cytotoxic drugs within 6 months before screening; Or those who received live attenuated vaccine within 1 month before screening;
4. Acute infection requiring treatment with intravenous antibiotics within 2 weeks before screening or current infection requiring antiinfective treatment;
5. Patients with clinically significant acute or chronic liver disease caused by non-HBV infection who were judged by the investigator to be unsuitable for the study;
6. A history of cirrhosis (e.g., the subject had a histopathological examination of the liver and reported cirrhosis, or had an endoscopic examination indicating varicose esophagus and fundus veins); Or currently confirmed or suspected decompensated cirrhosis, including but not limited to: hepatic encephalopathy, hepatorenal syndrome, hemorrhage of esophageal and fundus varices, spleen enlargement, ascites, etc.; Or there is evidence of progressive hepatic fibrosis;
7. Primary liver cancer; Serum AFP (AFP) is greater than 50 ㎍ / L (or 50 ng/mL) or imaging suggest possible malignant liver placeholder; Patients with other malignant tumors or a history of other malignant tumors within 5 years before screening (except cured basal cell or squamous cell carcinoma of the skin and cervical carcinoma in situ);
8. The presence of impaired gastrointestinal function or gastrointestinal disease that may affect oral drug absorption, such as severe gastrointestinal disease (peptic ulcer, erosive or atrophic gastritis), partial gastrectomy, and screening. Grade 2 gastrointestinal symptoms (e.g., nausea, vomiting, or diarrhea)；
9. Patients with severe circulatory, respiratory, urinary, blood, metabolic, immune, mental, nervous, renal and other diseases were judged by the researchers to be unsuitable for this study；
10. Patients with major trauma or major surgery within 3 months before screening; or plan to have surgery during the study;
11. Laboratory examination: platelet count < 90 x 10^9 / L; White blood cell count <3.0 x 10^9 / L; Neutrophils absolute value< 1.3 x 10^9 / L; Serum total bilirubin >2 x ULN. Albumin< 30 g/L; Creatinine clearance ≤ 60 mL/min or less; Prothrombin time international standardization ratio (INR) >1.5;
12. Hepatitis C antibody positive, AIDS antigen/antibody positive, treponema pallidum antibody positive and rapid plasma reagin test (RPR) positive;
13. Blood donation or blood loss ≥400 mL within 3 months prior to screening, or received blood transfusion; Or blood donation or blood loss ≥200 mL within 1 month before screening；
14. A history of continuous alcohol abuse (drinking > 14 alcohol units per week, defined as 1 alcohol unit for a 350ml bottle of beer, 120ml of wine, or 30ml of 40% spirits) within 3 years before screening;
15. A history of drug dependence or abuse;
16. Participants who participated in clinical trials of investigational drugs or medical devices within 3 months before screening and took investigational drugs or used medical devices;
17. Breastfeeding women or those who have a positive pregnancy test;
18. The investigator believes that there are other subjects who are not suitable for participating in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-08-24 (Actual)

PRIMARY OUTCOMES:
Serum HBV DNA | 12 or 24 weeks
  At the end of treatment, serum HBV DNA was lower than the lower limit of quantitative detection value (HBV DNA ≤ 20 IU/mL)percentage of subjects.

SECONDARY OUTCOMES:
Serum HBV DNA quantification | 12 or 24 weeks
  Changes in serum HBV DNA quantitative detection values from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- The first hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang C, Kong F, Gao H, Cai D, Zhang G, Ning Q, Zhong B, Liu Z, Su Z, Wu G, Hou J, Mao J, Zhang T, Wu W, Yan W, Yan X, Li G, Gao Y, Zhang G, Niu J. Safety and efficacy of GST-HG141, a novel HBV capsid assembly modulator, for the treatment of chronic hepatitis B patients with low-level viremia: a randomized, double-blind, placebo-controlled, multicenter phase II study. EClinicalMedicine. 2025 Aug 2;87:103400. doi: 10.1016/j.eclinm.2025.103400. eCollection 2025 Sep. PMID 40808966